CLINICAL TRIAL: NCT02709980
Title: Cognitive Behavior Therapy for Insomnia (CBT-I) in Persons With Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00062258
Record Dates: First submitted 2016-02-24; First posted 2016-03-16 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: TBI; Insomnia
Keywords: Brain Injury; Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep Education (Placebo Comparator): 6 sessions of sleep education.
  Interventions: Behavioral: Sleep Education
- Cognitive Behavior Therapy for Insomnia (Active Comparator): 6 sessions of cognitive behavioral therapy for insomnia (CBT-I).
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia

INTERVENTIONS:
Behavioral: Sleep Education — The sleep education intervention will parallel the CBT-I intervention in number, format (in-person) and length of sessions. It is intended to disseminate information about sleep including sleep hygiene information that is widely available. Subjects will be instructed to read and review 6 publications from the American Academy of Sleep Medicine; sessions will review the material to ensure complete access to the information.
  Arms: Sleep Education
Behavioral: Cognitive Behavior Therapy for Insomnia — Treatment will involve a standardized 6-session intervention, with demonstrated efficacy, that combines education and behavioral techniques to reduce insomnia. The core components include (1) education about sleep and insomnia, stimulus control, and sleep restriction (session 1); (2) sleep hygiene education (session 2); and 3) relaxation training, cognitive therapy, adherence monitoring, adjusting the recommended sleep-wake schedule, and addressing any problems in implementation (session 3-5). The final session will include a review of treatment content and relapse prevention.
  Arms: Cognitive Behavior Therapy for Insomnia

SUMMARY:
The current study seeks to evaluate cognitive behavior therapy for insomnia (CBT-I), a non-medication treatment, in recent TBI patients compared to a sleep education control intervention. Patients will participate in CBT-I treatment (or sleep education treatment) weekly for six weeks, and will have a 3-months follow-up visit in order to examine the efficacy and time course of treatment. In addition, participants will complete several self-report questionnaires in order to examine sleep and neuropsychiatric symptoms throughout treatment.

DETAILED DESCRIPTION:
Approximately 1.7 million people in the United States sustain a traumatic brain injury (TBI) every year due to various causes (falls, motor vehicle accidents, sports, work, etc.) [9] at an estimated combined cost of $110 billion made up of direct (e.g., medical) and indirect (e.g., lost productivity) costs [6]. Insomnia is one of the most common symptoms of traumatic brain injury (TBI). Sleep disturbance disrupts TBI recovery and increases the likelihood of developing neuropsychiatric symptoms, specifically putting TBI patients at enhanced risk for depressive and anxiety symptomatology. Standard pharmacological treatments used for managing insomnia are poor targets in this population, as they are vulnerable to medication side-effects. Very few non-pharmacological studies have been conducted to intervene on insomnia in this population. One such study hints at the effectiveness of cognitive behavioral therapy for insomnia (CBT-I). The current study seeks to evaluate CBT-I in recent TBI patients compared to a sleep education control intervention. Participants will wear a Fitbit and an Actiwatch to objectively evaluate sleep measures. Patients will participate in CBT-I treatment (or sleep education treatment) weekly for six weeks, and will have a 3-months follow-up visit in order to examine the efficacy and time course of treatment. In addition, participants will complete several self-report questionnaires in order to examine sleep and neuropsychiatric symptoms throughout treatment. This type of non-pharmacological multi-target therapy is much needed for persons with TBI, as they are at high risk of developing chronic neuropsychiatric sequelae but are vulnerable to medication side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Time duration since injury >3 and <60 months
* Report sleep problems for >1 month that developed after the TBI
* Insomnia Severity Index (ISI) score > or = 10
* Display sufficient cognitive capacity to provide informed consent (MoCA > 10)
* 18-65 years of age

Exclusion Criteria:

* Current alcohol or substance abuse/dependence
* Presence of other neurological disorders (e.g., multiple sclerosis, Parkinson's Disease)
* Presence of an untreated or unstable medical or psychiatric comorbid condition (e.g., major depressive disorder or psychotic disorder requiring admission). People using psychotropic medication, hypnotic or sedative medications may be included if they are on a stable dosage for the last 1 month prior to the study, if the dose remains stable throughout the study, and if the medication is judged to not interfere with the study outcomes.
* Currently on medications known to produce insomnia (e.g., stimulants)
* Cognitive communication difficulties or inability to speak English that would preclude study participation
* Sleep apnea (AHI >15) or previous diagnosis of. Study participants who use a continuous positive airway pressure (CPAP) device for sleep apnea will be eligible for participation if they are below the apnea/hypopnea cutoff while using CPAP and agree to use the device during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity | 5 months
  Insomnia severity will be operationalized as Sleep efficiency (an estimate of the amount of time spent sleeping relative to time in bed) = (Total time asleep) / (Time in Bed) x 100; sleep continuity (this will be derived from aggregating total time awake from the initial onset of sleep through the final awakening at the end of the sleep period); & total sleep time.

SECONDARY OUTCOMES:
Depressive Symptoms | 5 months
  Depression = Patients will complete psychometrically validated depressive symptoms questionnaires (e.g., Beck Depression Inventory, Patient Health Questionnaire - 9 item).
Anxiety Symptoms | 5 months
  Anxiety = Patients will complete psychometrically validated anxiety symptoms questionnaires (e.g., Beck Anxiety Inventory, Generalized Anxiety Disorder-7 item).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Buenaver, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided